CLINICAL TRIAL: NCT00480090
Title: A Phase II Study of Ara-C (Cytarabine) in Men With Androgen Independent Prostate Cancer
Acronym: SLAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLAP41206
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: Prostate; Androgen independent; Phase II; Second line; Androgen-independent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cytarabine (Experimental): eligible patients will receive cytarabine, starting at 075g/m2 and escalating to a maximum of 1.25g/m2, BID IV for 2 days every three weeks for 6 or more cycles if tolerated.
  Interventions: Drug: Cytarabine

INTERVENTIONS:
Drug: Cytarabine — Initially given at 1g/m2 bid for 2 days every 3 weeks over 2 hours. The dose will be escalated: level 1 - 1.25g/m2, level 2, 1.5g/m2.

SUMMARY:
This is a single-arm, open label phase II trial of the investigational agent, Ara-C (cytarabine), in patients diagnosed with hormone refractory prostate cancer whose disease has progressed on or deemed not suitable for standard chemotherapy with docetaxel. Ara-C appears to inhibit DNA synthesis and is cytotoxic to a wide variety of mammalian cells. Recent discoveries have suggested the role of gene fusions in the ETS family of transcription factors as important for the development of prostate cancer. Ara-C appears to block ETS genes, suggesting that it is worthwhile to explore Ara-C as a potential new treatment for patients with hormone refractory prostate cancer given that there is no standard of care for the proposed patient population. In this study, Ara-C will be administered intravenously for 2 days every 3 weeks (1 cycle). Treatment will be for 6 cycles if tolerated and may be continued in patients who are responding and do not have severe toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven prostate cancer or clinical picture consistent with metastatic prostate cancer with high level of serum PSA (> 20ng/ml)
* At least 4 weeks after docetaxel treatment and have at least 2 consecutive rising PSAs measured at least 2 weeks apart
* Progression on or intolerance of docetaxel chemotherapy
* ECOG performance status ≤ 2
* Adequate organ and marrow function

Exclusion Criteria:

* Prior treatment with cytarabine
* Receiving any other investigational or anticancer agents
* Uncontrolled intercurrent illness
* Active malignancy at any other site excluding squamous cell or basal cell carcinomas of the skin
* Radiotherapy within the past 4 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
PSA response | 50% decline in PSA from baseline, confirmed by a second measurement ≥3 weeks later
  PSA levels will be collected at screening, baseline, 2 weeks following study termination, and upon followup to determine PSA level response to treatment.

SECONDARY OUTCOMES:
Pain response | Baseline median PPI with no concomitant increase in analgesic score/pain
  Patients will complete Present Pain Intensity (PPI) scale a baseline, every three weeks during treatment and at the end of study.
QOL response | Baseline to two measurements obtained at least three weeks apart
  Quality of Life (QOL) will be assessed with the Functional Assessment of Cancer Therapy - Prostate questionnaire, self administered by patients.
PSA progression free survival | Baseline and the date of PSA progression or the date of death due to prostate cancer, whichever occurs first.
  Time between randomization date and the date of PSA progression (>25% increase from baseline) or the date of death due to prostate cancer, whichever occurs first.
Measurable disease response | Every 3 cycles (9 weeks)
  Radiological measurement of effect. Measurement at baseline, and every 3 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Joshua, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada